CLINICAL TRIAL: NCT00338715
Title: A Randomized Controlled Trial of Prophylactic Pulmonary Vein Isolation as Adjunct to Coronary Artery Bypass Grafting
Brief Title: Effectiveness of Pulmonary Vein Isolation in Prevention of Atrial Fibrillation Following Heart Bypass Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Dr. Bob Kiaii, London Health Sciences Centre, University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R-06-035; 11973
Record Dates: First submitted 2006-06-19; First posted 2006-06-20 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2011-02

CONDITIONS: Atrial Fibrillation
Keywords: Effectiveness; Pulmonary Vein Isolation Procedure; Coronary Artery Bypass Surgery; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Prophylactic Pulmonary Vein Isolation in Addition to CABG for the prevention of postoperative Atrial Fibrillation
  Interventions: Device: PVI with Medtronic's Cardioblate BP2 radiofrequency catheter

INTERVENTIONS:
Device: PVI with Medtronic's Cardioblate BP2 radiofrequency catheter — Ablation of the right and left pulmonary veins
  Other Names: Medtronic's Cardioblate BP2 radiofrequency catheter

SUMMARY:
Atrial fibrillation (AF) is an irregular heart rhythm that occurs in 30% to 40% of patients following heart surgery. This irregular heart rhythm, although often self-limiting, can be cause for concern. AF is associated with a two-fold increase in patient complications and mortality after heart surgery. During AF, the heart muscle does not contract properly causing the blood flow through the heart to slow down potentially forming clots. A clot may then enter the blood stream and be carried to the brain, possibly causing a stroke. Patients in persistent AF require blood thinners to prevent strokes, and this carries its own bleeding risks especially in elderly patients.

Patients in AF after heart surgery spend twice as many days in the intensive care unit and 3 to 4 more days in the hospital, hence the impact on hospital resources is quite significant. Various medications are used to prevent AF after heart surgery but they are unable to completely prevent this complication and the medications have associated side effects. In an effort to optimize the care of heart surgery patients, strategies set on eliminating the onset of AF after surgery, as opposed to trying to control AF with less than effective medications, is a necessity.

We are proposing a study to determine if isolating the misfiring areas that cause AF at the time of bypass surgery in high-risk patients will decrease the occurrence of AF following heart surgery. Consenting patients will be randomized to one of two groups. Group 1 will undergo bypass surgery plus the additional procedure of pulmonary vein isolation and Group 2 will undergo bypass surgery only, without the additional procedure. Four staff cardiac surgeons at the London Health Sciences Centre will perform all surgeries. Patients will be seen postoperatively every six months and will be followed for a two-year period. The occurrence of AF will be recorded as well as other complications and lengths of hospital stay. We predict that the group with the additional pulmonary vein isolation procedure to prevent AF will have a much lower occurrence of this complication. If this is found to be beneficial, this will significantly decrease the complications and mortality associated with heart surgery. This will have a profound effect in the delivery of care to patients with coronary artery disease and other forms of heart disease.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is a well recognized postoperative complication associated with cardiac surgery occurring in approximately 30% to 40% of patients. AF occurs most frequently within 24 to 72 hours after surgery. Even though postoperative AF is often a short-lived, self-limiting complication, it is associated with a two-fold increase in cardiovascular mortality and morbidity. Patients are often symptomatic due to irregular and/or rapid ventricular rates and complain of palpitations, anxiety, and diminished physical capacity. Postoperative AF is associated with increased incidence of other complications and increased hospital length of stay and overall costs. Patients may also develop congestive heart failure and hemodynamic instability as a result of this complication. As a result of stasis in the left atrium, the risk of thromboembolic complications is increased and the incidence of postoperative stroke is increased. Patients with persistent AF have a 13-fold higher hospital stroke rate than patients without persistent AF. Further morbidity is added in patients requiring anticoagulation if AF lasts greater than 48 hours. Elderly patients requiring anticoagulation have a significantly increased risk of hemorrhagic complications. The incidence of ventricular arrhythmias is also increased in patients in whom AF develops after cardiac operations.

Postoperative AF has an immense impact on both the cardiac surgery patient and hospital resources. One study determined that patients developing AF after cardiac surgery spend about twice as many days in the Intensive Care Unit as patients without AF, and their hospital stay is extended by 3-4 days.Strategies aimed at preventing postoperative AF are necessary to optimize the postoperative care of patients undergoing open heart operations. A large number of clinical trials have evaluated the effectiveness of various pharmacologic modalities in decreasing rates of AF following cardiac surgery. A recent meta-analysis demonstrated that beta blockers, sotalol and amiodarone all reduce the risk of postoperative AF with no marked difference between them. However, neither agent completely eliminated the occurrence of postoperative AF. In the largest available beta blocker prevention trial, metoprolol decreased the prevalence of postoperative AF from 39% to 31%.

The mechanism of AF following cardiac surgery is not well understood, but possible etiologies include rapid firing from an ectopic focus and multiple reentrant circuits within the atria to propagate this rhythm. It has been discovered that in chronic and paroxysmal AF, the pulmonary veins and the surrounding ostial areas frequently contain focal triggers or re-entrant circuits critical to the initiation of AF. In a study of 45 patients with frequent episodes of AF refractory to drug therapy, 94% of ectopic beats responsible for instigating AF were located in the pulmonary veins. Studies have shown that these foci are responsive to radiofrequency ablation. Although it has never been used in the prevention of postoperative AF, circumferential pulmonary vein ablation (CPVA) is a technique that has shown much success in the treatment of AF. In CPVA, radiofrequency lesions are created around the ostia of each pulmonary vein, with the aim to electrically isolate these veins from the left atrium. In one study, 26 patients with resistant AF were treated with CPVA and 64% had sinus rhythm restoration during ablation. In addition, 85% of patients were free of AF at 9 months, with 62% no longer requiring antiarrhythmic drugs and 23% taking drugs that had been ineffective before ablation. Radiofrequency pulmonary vein isolation with electro-anatomic guidance is a safe and effective treatment of AF.

Recently, Medtronic has developed the Cardioblate® BP and BP 2 Surgical Ablation System devices (Minneapolis, MN) to perform pulmonary vein isolation to treat AF. Vichol et al have demonstrated a mean ablation time of 15.2 seconds per lesion with the use of this device.

It is clearly evident that postoperative AF increases morbidity, length of hospital stay, and costs associated with surgical coronary artery revascularization. The current prophylactic agents are not completely effective at eliminating the occurrence of postoperative AF. It has been shown that pulmonary vein isolation is an effective method of treating patients with chronic AF. We propose a study to determine if performing pulmonary vein isolation with the Cardioblate® BP 2 as an adjunct in those patients undergoing routine coronary artery bypass surgery, who are at increased risk of developing postoperative AF, will significantly reduce the occurrence of this complication.

If pulmonary vein isolation is found to considerably decrease the incidence of postoperative AF, the associated morbidity will also be decreased. This will have a very profound effect in the delivery of care to patients with ischemic heart disease.

Study Question/Purpose:

In patients at an increased risk of developing postoperative atrial fibrillation following coronary artery bypass grafting, does pulmonary vein isolation with Cardioblate® BP 2 result in a decreased incidence of postoperative atrial fibrillation when compared to those patients that do not have this adjunct procedure?

Hypothesis:

Pulmonary vein isolation with Cardioblate® BP 2 will reduce the incidence of postoperative atrial fibrillation in patients undergoing coronary artery bypass grafting who are at an increased risk of developing postoperative atrial fibrillation.

Sample Size A sample size of 79 patients per group was calculated to detect a reduction in incidence of postoperative atrial fibrillation from 40% to 20% using a two-sided α = 0.05 and a power of 80%.

Blinding-The patients, outcome assessors, and data analysts will be blinded to which group the patients belong. Allocation concealment will be practiced and the randomization scheme will not be revealed. Due to the nature of the intervention, it is not possible to blind the surgeon performing the operation.

Trial Implementation

After randomization is complete, the baseline demographic characteristics of all patients will be recorded. Those patients randomized to the control group will undergo coronary bypass grafting with cardiopulmonary bypass. Those patients randomized to the experimental group will undergo coronary artery bypass grafting with cardiopulmonary bypass (CABG) and pulmonary vein isolation (PVI). Medtronic's Cardioblate® BP 2 will be used for the pulmonary vein isolation. The following will take place for each patient:

1. Will be transferred to the Cardiac Surgery Recovery Unit following surgery
2. Cardiac rhythm will be monitored with telemetry in the CSRU and on the floor until discharge home
3. All arrhythmias will be documented with regards to onset, duration, and immediate management - will be recorded by research assistant
4. All patients will be started on a beta blocker on POD #1 and will continue for minimum 2 years if tolerable - will be discontinued if any adverse effect (i.e., heart block, decreased cardiac output, allergic reaction)
5. All medications will be documented
6. After discharge home, all complications and readmissions will be documented (i.e., development of atrial fibrillation or other arrhythmia)
7. Documentation of those patients requiring anticoagulation for persistent atrial fibrillation and duration and complications related to anticoagulation
8. Follow-up of patients by surgeons, cardiologist and research assistant with ECG every 6 months for 2 years - patients will be asked to fill out questionnaire at each visit that may elicit any symptoms related to arrhythmias Outcomes Statistical Analysis All outcomes will be analyzed by a biostatistician blinded to allocation groups using the intention to treat principle. The primary purpose of the data analyses is to determine whether pulmonary vein isolation reduces the incidence of postoperative atrial fibrillation in patients undergoing coronary artery bypass grafting who are at high risk of developing postoperative atrial fibrillation. The primary outcome will be compared between both groups with the Chi-square test. All patients will be accounted for and we will aim for 100% follow-up for all patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (Age>=18) undergoing elective coronary artery bypass grafting with cardiopulmonary bypass by 4 surgeons at the London Health Sciences Centre
* Patients at high risk of developing postoperative atrial fibrillation--patients are required to meet one or more of the following criteria:
* Age >=65
* Ejection Fraction <50% or Left Ventricle Grade of 2-3
* Diabetes Mellitus (independent of type of management)

Exclusion Criteria:

* Any documented prior history of atrial fibrillation (paroxysmal/chronic)
* Contraindication to Beta Blockers
* Severe COPD with intolerance to Beta Blockers
* Concomitant non-CABG procedure
* Enrollment in another RCT
* Inability to obtain informed consent
* Patients' inability to attend follow-up visits
* Grade IV left ventricle (EF <20%)
* Redo CABG procedure
* Off-pump coronary artery bypass surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2006-07; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative atrial fibrillation as documented on telemetry/ECG for >=30 minutes while in hospital or AF requiring immediate intervention ie.cardioversion | while in hospital

SECONDARY OUTCOMES:
Composite endpoint of perioperative death +/- one of 10 major complications. | while in hospital and within 30 days of discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Bob Kiaii, MD, FRCSC, Principal Investigator — Department of Cardiac Surgery, University of Western Ontario and the London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, University Hospital, London, Ontario, Canada

REFERENCES:
- [Background] Crystal E, Connolly SJ, Sleik K, Ginger TJ, Yusuf S. Interventions on prevention of postoperative atrial fibrillation in patients undergoing heart surgery: a meta-analysis. Circulation. 2002 Jul 2;106(1):75-80. doi: 10.1161/01.cir.0000021113.44111.3e. PMID 12093773
- [Background] DiDomenico RJ, Massad MG. Pharmacologic strategies for prevention of atrial fibrillation after open heart surgery. Ann Thorac Surg. 2005 Feb;79(2):728-40. doi: 10.1016/j.athoracsur.2004.03.037. PMID 15680883
- [Background] Onalan O, Lashevsky I, Crystal E. Prophylaxis and management of postoperative atrial fibrillation. Curr Cardiol Rep. 2005 Sep;7(5):382-90. doi: 10.1007/s11886-005-0093-4. PMID 16105495
- [Background] Crystal E, Healey J, Connolly SJ. Atrial fibrillation after cardiac surgery: update on the evidence on the available prophylactic interventions. Card Electrophysiol Rev. 2003 Jun;7(2):189-92. doi: 10.1023/a:1027432104518. PMID 14618049
- [Background] Crystal E, Garfinkle MS, Connolly SS, Ginger TT, Sleik K, Yusuf SS. Interventions for preventing post-operative atrial fibrillation in patients undergoing heart surgery. Cochrane Database Syst Rev. 2004 Oct 18;(4):CD003611. doi: 10.1002/14651858.CD003611.pub2. PMID 15495059
- [Background] Elahi M, Hadjinikolaou L, Galinanes M. Incidence and clinical consequences of atrial fibrillation within 1 year of first-time isolated coronary bypass surgery. Circulation. 2003 Sep 9;108 Suppl 1:II207-12. doi: 10.1161/01.cir.0000089188.45285.fd. PMID 12970234
- [Background] Vicol C, Eifert S, Kur F, Reichart B. Minimally invasive off-pump pulmonary vein isolation to treat paroxysmal atrial fibrillation. Thorac Cardiovasc Surg. 2005 Jun;53(3):176-8. doi: 10.1055/s-2005-837527. PMID 15926099
- [Background] Ishii Y, Schuessler RB, Gaynor SL, Yamada K, Fu AS, Boineau JP, Damiano RJ Jr. Inflammation of atrium after cardiac surgery is associated with inhomogeneity of atrial conduction and atrial fibrillation. Circulation. 2005 Jun 7;111(22):2881-8. doi: 10.1161/CIRCULATIONAHA.104.475194. Epub 2005 May 31. PMID 15927979
- [Background] Stamou SC, Dangas G, Hill PC, Pfister AJ, Dullum MK, Boyce SW, Bafi AS, Garcia JM, Corso PJ. Atrial fibrillation after beating heart surgery. Am J Cardiol. 2000 Jul 1;86(1):64-7. doi: 10.1016/s0002-9149(00)00829-8. PMID 10867094